CLINICAL TRIAL: NCT01830660
Title: A Phase I, Randomized, Placebo-controlled, Ascending Single And Multiple Oral Dose Study To Investigate Safety, Tolerability, Pharmacokinetics, And Pharmacodynamics Of Hetrombopag Olamine (SHR8735 Olamine) In Healthy Subjects
Brief Title: A Phase I Study of Hetrombopag Olamine in Healthy Adult Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SHR-TPOP1
Record Dates: First submitted 2012-12-25; First posted 2013-04-12 (Estimated); Last update posted 2015-04-06 (Estimated); Status verified 2013-04

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- hetrombopag (Experimental): hetrombopag either at 2.5,5,10,20,30 or 40mg, p.o. once daily
  Interventions: Drug: Hetrombopag Olamine Tablets
- placebo (Placebo Comparator): Subjects will be randomized (5:1 eltrombopag : placebo) to receive either eltrombopag or placebo.
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Hetrombopag Olamine Tablets
  Arms: hetrombopag
Drug: placebo
  Arms: placebo

SUMMARY:
Hetrombopag Olamine made by Jiangsu Hengrui Medicine co Ltd. has shown an effect of increasing platelet count in animal and human. This study is designed in dose escalation fashion to evaluate safety, pharmacokinetics and efficacy of Hetrombopag Olamine.

DETAILED DESCRIPTION:
1. To evaluate safety and tolerability of Hetrombopag Olamine.
2. To investigate pharmacokinetics of Hetrombopag Olamine Under fasting conditions.
3. To obtain pharmacodynamics information of Hetrombopag Olamine on platelet count elevation in healthy volunteers.
4. To determine preliminary regimen for phase II study.

ELIGIBILITY:
Inclusion Criteria:

1. Subject must be adequately informed of the nature and risks of the study, able to understand the risks associated with the study, and are willing to provide written informed consent prior to screening.
2. Must be a healthy male between the ages of 18 to 45 years, inclusive.
3. Must have a BMI between 19 to 28 kg/m2, inclusive and a total body weight ≥50 kg.
4. Platelet counts must be within the normal range.
5. Subjects must be free of any clinically significant disease based on medical history and physical examination.
6. Clinical laboratory tests (complete blood count [CBC], blood chemistries, and urinalysis) must be within the normal limits or clinically acceptable.
7. Must be nonsmokers, defined as not having smoked tobacco or used chewing tobacco or nicotine.
8. Subjects of reproductive potential with partners who are women of childbearing potential, will be instructed to, and must be willing to practice a highly effective method of birth control for the duration of the study and continuing 6 months after discontinuing treatment with the investigational product.

Exclusion Criteria:

1. History of hypersensitivity to hetrombopag olamine or its components.
2. History or presence of significant cardiovascular deficient, pulmonary, hepatic, gallbladder or biliary tract, renal, hematological, gastrointestinal, endocrine, immunological, dermatological, neurological, or psychiatric disease, or any other condition known to interfere with the absorption, distribution, metabolism, or excretion of drugs.
3. History of deep vein thrombosis, or any other thromboembolic event.
4. History or presence of conditions that may place the subject at increased risk as determined by the investigator.
5. History of thrombocytopenia or bleeding due to abnormal platelet number or function.
6. History of platelet clumping that prevents reliable measurement of platelet counts.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 96 (Estimated)
Dates: Start 2012-04; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Change in platelet count above baseline(%)on Day1,3,5,8,10,12,15,17,19,22,25,28 after dosing | up to 4 weeks
Composite pharmacokinetic (PK) parameters of eltrombopag following a single dose of eltrombopag | For 5 days

SECONDARY OUTCOMES:
Adverse events | up to 4 weeks
Change in vital signs | up to 4 weeks
Change in clinical laboratory parameters | up to 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Maozhi Liang, Dr, Principal Investigator — West China Hospital
Locations (1):
- West China Hospital, Sichuan University, Chengdu, Sichuan, China